CLINICAL TRIAL: NCT03044665
Title: RAndomized Comparison of Efficacy and Safety of Lipid-lowerING With Statin Monotherapy Versus Statin/Ezetimibe Combination for High-risk Cardiovascular Diseases (RACING Trial)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-1025
Record Dates: First submitted 2017-02-01; First posted 2017-02-07 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Diseases; Cerebrovascular Disease; Peripheral Atherosclerotic Disease
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-intensity statin monotherapy (Active Comparator): Statin monotherapy
  Interventions: Drug: Rosuvastatin
- Statin plus ezetimibe combination therapy (Experimental): Statin plus ezetimibe combination therapy
  Interventions: Drug: Rosuvastatin plus ezetimibe

INTERVENTIONS:
Drug: Rosuvastatin — Subjects will start rosuvastatin 20 mg a day irrespective of previous lipid-lowering treatment or LDL-cholesterol level as current US guideline.
  Arms: High-intensity statin monotherapy
Drug: Rosuvastatin plus ezetimibe — Subjects will start single combination pill of rosuvastatin 10 mg plus ezetimibe 10 mg a day irrespective of previous lipid-lowering treatment or LDL-cholesterol level.
  Arms: Statin plus ezetimibe combination therapy

SUMMARY:
The clinical efficacy of LDL-lowering therapy have been proven with strong evidences and more emphasized. However, there are also growing concerns that high-intensity statin would be related to increased risk of adverse effects. In addition, there was an inconsistency of efficacy of statin according to ethnic population. Asian population showed more profound LDL reduction not only from high potent statin but from moderate to low potent statin. Conventional strategies for lowering LDL-cholesterol was focused on statins, therefore doubling of previously described dose of statin would be common way in patients with inadequate lowering LDL-cholesterol level. Additive ezetimibe will also an alternative strategy not only to lower LDL-cholesterol level and also to reduce the need of dosage of high-intensity statin to fulfill sufficient LDL-cholesterol lowering effect. We will evaluate whether additive ezetimibe with rosuvastatin will have comparable clinical efficacy in terms of clinical outcomes and goal attainment of LDL-C compared to rosuvastatin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-80 years
* Documented CVD (cardiovascular disease), previous MI(Myocardial Infarction), ACS (Acute Coronary Syndrome), coronary revascularization and other arterial revascularization procedures, ischemic stroke, or PAD (peripheral artery disease)

Exclusion Criteria:

* Active liver disease or persistent unexplained serum AST or ALT elevation more than 2 times the upper limit of normal range
* Allergy or hypersensitivity to any statin or ezetimibe
* Solid organ transplantation recipient
* History of any adverse drug reaction requiring discontinuation of statin
* Pregnant women, women with potential childbearing, or lactating women
* Life expectancy less than 3 years
* Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator
* Inability to understand or read the informed content

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3780 (Estimated)
Dates: Start 2017-03-15 (Actual); Primary Completion 2022-01-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular death | Clinical status including medication and clinical events will be evaluated at 2 months.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Composite of cardiovascular death | Clinical status including medication and clinical events will be evaluated at 6 months.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Composite of cardiovascular death | Clinical status including medication and clinical events will be evaluated at every years until 3 years.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Major cardiovascular event | Clinical status including medication and clinical events will be evaluated at 2 months.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Major cardiovascular event | Clinical status including medication and clinical events will be evaluated at 6 months.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Major cardiovascular event | Clinical status including medication and clinical events will be evaluated at every years until 3 years.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Composite of nonfatal stroke | Clinical status including medication and clinical events will be evaluated at 2 months.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Composite of nonfatal stroke | Clinical status including medication and clinical events will be evaluated at 6 months.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
Composite of nonfatal stroke | Clinical status including medication and clinical events will be evaluated at every years until 3 years.
  Composite of cardiovascular death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)

SECONDARY OUTCOMES:
Clinical efficacy of lipid lowering treatment | 3years
  1. The proportion of participants whose LDL cholesterol is lower than 70mg/dL (1,2,3 years after enrollment)
  2. Composite of all death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
  3. Statin discontinuation or dose-reduction caused by intolerance
  4. new-onset DM, muscle-related adverse events, gastrointestinal symptom, gallbladder-related event, major bleeding, cancer, new-onset neurocognitive disorder, cataract surgery
Clinical safety of lipid lowering treatment | 3years
  1. The proportion of participants whose LDL cholesterol is lower than 70mg/dL (1,2,3 years after enrollment)
  2. Composite of all death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
  3. Statin discontinuation or dose-reduction caused by intolerance
  4. new-onset DM, muscle-related adverse events, gastrointestinal symptom, gallbladder-related event, major bleeding, cancer, new-onset neurocognitive disorder, cataract surgery
statin discontinuation and intolerance | 3years
  1. The proportion of participants whose LDL cholesterol is lower than 70mg/dL (1,2,3 years after enrollment)
  2. Composite of all death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
  3. Statin discontinuation or dose-reduction caused by intolerance
  4. new-onset DM, muscle-related adverse events, gastrointestinal symptom, gallbladder-related event, major bleeding, cancer, new-onset neurocognitive disorder, cataract surgery
Clinical adverse events | 3years
  1. The proportion of participants whose LDL cholesterol is lower than 70mg/dL (1,2,3 years after enrollment)
  2. Composite of all death, major cardiovascular event, nonfatal stroke (Major cardiovascular event include any coronary or peripheral revascularization and hospitalization for any cardiovascular events including ischemic heart disease, heart failure, peripheral arterial disease.)
  3. Statin discontinuation or dose-reduction caused by intolerance
  4. new-onset DM, muscle-related adverse events, gastrointestinal symptom, gallbladder-related event, major bleeding, cancer, new-onset neurocognitive disorder, cataract surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee JH, Ahn SG, Jeon HS, Lee JW, Youn YJ, Lee YJ, Lee SJ, Hong SJ, Ahn CM, Ko YG, Kim JS, Choi D, Hong MK, Jang Y, Kim BK. Remnant cholesterol as a residual risk in atherosclerotic cardiovascular disease patients under statin-based lipid-lowering therapy: A post hoc analysis of the RACING trial. J Clin Lipidol. 2024 Nov-Dec;18(6):e905-e914. doi: 10.1016/j.jacl.2024.07.005. Epub 2024 Jul 27. PMID 39322526
- [Derived] Kim BG, Lee SJ, Lee YJ, You SC, Hong SJ, Yun KH, Hong BK, Heo JH, Rha SW, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y, Cho YH, Kim JS. Effect of moderate-intensity statin with ezetimibe combination vs. high-intensity statin therapy according to sex in patients with atherosclerosis. Sci Rep. 2023 Nov 17;13(1):20157. doi: 10.1038/s41598-023-47505-x. PMID 37978309
- [Derived] Lee SJ, Cha JJ, Choi WG, Lee WS, Jeong JO, Choi S, Cho YH, Park W, Yoon CH, Lee YJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y, Hong SJ, Kim JS; RACING Investigators. Moderate-Intensity Statin With Ezetimibe Combination Therapy vs High-Intensity Statin Monotherapy in Patients at Very High Risk of Atherosclerotic Cardiovascular Disease: A Post Hoc Analysis From the RACING Randomized Clinical Trial. JAMA Cardiol. 2023 Sep 1;8(9):853-858. doi: 10.1001/jamacardio.2023.2222. PMID 37531130
- [Derived] Park JI, Lee SJ, Hong BK, Cho YH, Shin WY, Lim SW, Kang WC, Park Y, Lee SY, Lee YJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y, Kim JS; RACING investigators. Efficacy and safety of moderate-intensity statin with ezetimibe combination therapy in patients after percutaneous coronary intervention: a post-hoc analysis of the RACING trial. EClinicalMedicine. 2023 Apr 4;58:101933. doi: 10.1016/j.eclinm.2023.101933. eCollection 2023 Apr. PMID 37090440
- [Derived] Lee SH, Lee YJ, Heo JH, Hur SH, Choi HH, Kim KJ, Kim JH, Park KH, Lee JH, Choi YJ, Lee SJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y, Kim JS. Combination Moderate-Intensity Statin and Ezetimibe Therapy for Elderly Patients With Atherosclerosis. J Am Coll Cardiol. 2023 Apr 11;81(14):1339-1349. doi: 10.1016/j.jacc.2023.02.007. PMID 37019580
- [Derived] Lee YJ, Cho JY, You SC, Lee YH, Yun KH, Cho YH, Shin WY, Im SW, Kang WC, Park Y, Lee SY, Lee SJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y, Kim JS. Moderate-intensity statin with ezetimibe vs. high-intensity statin in patients with diabetes and atherosclerotic cardiovascular disease in the RACING trial. Eur Heart J. 2023 Mar 14;44(11):972-983. doi: 10.1093/eurheartj/ehac709. PMID 36529993
- [Derived] Kim BK, Hong SJ, Lee YJ, Hong SJ, Yun KH, Hong BK, Heo JH, Rha SW, Cho YH, Lee SJ, Ahn CM, Kim JS, Ko YG, Choi D, Jang Y, Hong MK; RACING investigators. Long-term efficacy and safety of moderate-intensity statin with ezetimibe combination therapy versus high-intensity statin monotherapy in patients with atherosclerotic cardiovascular disease (RACING): a randomised, open-label, non-inferiority trial. Lancet. 2022 Jul 30;400(10349):380-390. doi: 10.1016/S0140-6736(22)00916-3. Epub 2022 Jul 18. PMID 35863366